CLINICAL TRIAL: NCT05580406
Title: Outreach to Reduce Depression Disparities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: Henry Ford Health System (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12874
Record Dates: First submitted 2022-10-11; First posted 2022-10-14 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2024-10

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Usual Care (No Intervention): Participants assigned to usual care will not receive outreach messages (online or via telephone) by study staff.
- Outreach Messaging (Experimental): Participants in the outreach messaging arm will receive messages via online secure message system (embedded within the health care record) and/or telephone.
  Interventions: Behavioral: Outreach messaging

INTERVENTIONS:
Behavioral: Outreach messaging — Participants will receive outreach messages via health care system secure messaging and/or phone following a new diagnosis of depression made in primary care if the participant has failed to initiate treatment (pharmacotherapy or psychotherapy) within 30 days of new diagnosis.
  Arms: Outreach Messaging

SUMMARY:
Previous research by Mental Health Research Network (MHRN) investigators and others demonstrates that online messaging and other telehealth technologies can effectively and efficiently address premature discontinuation of depression treatment. These interventions, however, have focused on adherence after treatment initiation and have been tested primarily in non-Hispanic white populations. Less is known about the acceptability and effectiveness of different communication modalities (online messaging, mailed letters, telephone) among racial and ethnic minority populations. Implementation of electronic-Health (eHealth) technologies must take care not to exacerbate health disparities.

This clinical trial involves a pilot trial to evaluate a population-based outreach program to improve rates of depression treatment initiation among traditionally underserved racial and ethnic groups. This pilot work intends to inform a subsequent full-scale pragmatic trial to examine impact on health disparities.

ELIGIBILITY:
Inclusion Criteria:

* New diagnosis of major depressive disorder or dysthymic disorder at a primary care visit ("new" defined as no depression diagnosis, psychotherapy visit or filled antidepressant prescription in the prior year)
* Continuously enrolled in the participating health system for 365 days prior to the eligible diagnosis (to assure capture of prior diagnoses or treatments)
* Patients Health Questionnaire-9 (PHQ-9) depression score of 10 or more within 14 days before to 7 days after the eligible diagnosis
* No filled prescription for any antidepressant medication OR psychotherapy visit attended within 30 days of the eligible diagnosis*
* No recorded PHQ-9 depression score less than 5 since the eligible diagnosis
* At least 18 years of age or older

Exclusion Criteria:

* Diagnosis of schizophrenia or bipolar disorder in the prior 2 years
* Not registered to use Electronic Health Record (EHR) patient portal
* Previously requested to not be contacted for research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 322 (Actual)
Dates: Start 2023-04-13 (Actual); Primary Completion 2024-12-10 (Actual); Study Completion 2024-12-10 (Actual)

PRIMARY OUTCOMES:
Initiation of formal depression treatment | within 60 days of randomization
  Defined as either at least one filled prescription for any antidepressant medication or attending at least one individual psychotherapy visit.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Kaiser Permanente, Hawaii Market, Honolulu, Hawaii
  - Henry Ford Health, Detroit, Michigan

IPD SHARING:
Plan to Share IPD: No